CLINICAL TRIAL: NCT02852486
Title: Pilot Study of Imatinib Discontinuation in Patients With Chronic Myeloid Leukemia With Deep Molecular Response - Evaluation of Pioglitazone in Treatment-free Remission (EDI-PIO)
Brief Title: Study of Imatinib Discontinuation in Chronic Myeloid Leukemia With Deep Molecular Response
Acronym: EDI-PIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Katia B. B. Pagnano, Hematologist, Hemocentro-Unicamp, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EDI-PIO-UNICAMP
Record Dates: First submitted 2016-07-09; First posted 2016-08-02 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Chronic Myeloid
Keywords: BCR-ABL Positive; Leukemia, Chronic Myeloid; Imatinib; Pioglitazone
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Pioglitazone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental): Pioglitazone will be given 30 mg/day, orally, for 3 months, before imatinib discontinuation
  Interventions: Drug: Pioglitazone 30 Mg Oral Tablet; Other: imatinib discontinuation

INTERVENTIONS:
Drug: Pioglitazone 30 Mg Oral Tablet — 30 mg/day, orally, for 3 months, before imatinib discontinuation
  Other Names: cloridrato de pioglitazona 30mg EMS S/A, Brasil
Other: imatinib discontinuation — imatinib discontinuation after 3 months of pioglitazone

SUMMARY:
The purpose of this study is to evaluate treatment-free remission after imatinib discontinuation in patients with chronic myeloid leukemia with deep molecular response. Before discontinuation, patients will receive pioglitazone associated with imatinib during 3 months.

DETAILED DESCRIPTION:
Treatment of chronic myeloid leucemia (CML) with tyrosine kinase inhibitors (TKIs) changed dramatically the prognosis of CML, with high rates of cytogenetic and molecular remission and increase of overall and progression-free survival. However, the long-term treatment of CML has a high cost to the health system, due to the price of these drugs and the need for continued use. In addition, chronic adverse effects may compromise the quality of life of patients. Discontinuation trials of TKIs have been developed in order to identify groups of patients who may benefit from treatment discontinuation if they have obtained deeper molecular responses.The primary objective of this study is to evaluate treatment free remission (TFR) after imatinib discontinuation in patients treated for more than 3 years with imatinib and with deep molecular response stable for two years (defined in the present study as a molecular response of 4.5 log reduction in breakpoint cluster region (BCR)-Abelson murine leukemia viral oncogene homolog 1(ABL) transcripts levels according to the international scale (MR 4.5; BCR-ABL/ABL ratio < or = 0.0032%). Patients with these criteria will receive pioglitazone for 3 months concomitant with imatinib, prior to discontinuation. After imatinib discontinuation, patients will be evaluated by molecular assessment of BCR-ABL transcripts levels by quantitative real time polymerase chain reaction (RQ-PCR) monthly during the first year, every 2 months in the second year and then every 3 months. The criteria for restarting treatment will be the loss of major molecular response (MMR), documented by a single RQ-PCR test > 0.1%, or confirmed loss of 4 log reduction molecular response (MR4.0), by 2 consecutive RQ-PCR tests > 0.01%.

ELIGIBILITY:
Inclusion Criteria:

* CML in chronic phase
* treatment with imatinib for 3 or more years
* MR4.5 (RQ-PCR< ou =0.0032%) confirmed by 4 RQ-PCR tests for BCR-ABL in the last 2 years (2 tests within the last 6 months)
* Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 reference level
* Bilirubins ≤ 1.5 reference level
* Contraceptive precautions for women

Exclusion Criteria:

* Patients less than 18 years
* Severe organ disfunction (liver or kidney)
* Severe cardiovascular disease: grade I-IV from New York Heart Association (NYHA) or acute myocardial infarction in the last six months, symptomatic arrhythmias
* Fluid retention grade 3 or 4
* Osteoporosis in treatment
* Patients with previous CML in accelerated or blast phase or blast or Philadelphia positive (Ph+) acute lymphoid leukemia (ALL)
* BCR-ABL mutations related to resistance
* Previous allogeneic bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Treatment-free remission after imatinib discontinuation | Through study completion (five years)
  Treatment-free remission time after imatinib discontinuation in patients with CML treated with pioglitazone for 3 months before imatinib discontinuation. Calculated from the date of imatinib discontinuation until imatinib reintroduction
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  assessment of number of participants with treatment-related adverse events as assessed by CTCAE v4.0 during the 3 months of treatment with imatinib and pioglitazone

SECONDARY OUTCOMES:
proportion of patients with MMR, MR4.0, MR4.5 | 3, 6 and 12 months
  Proportion of patients with MMR, MR4.0 and MR4.5 at 3, 6 and 12 months after imatinib discontinuation
Time from imatinib discontinuation until loss of MMR | Through study completion (five years)
  Time measured from the date of imatinib discontinuation until the date of loss of MMR, in days
Rate of loss of complete cytogenetic response | Through study completion (five years)
  % of patients who lost complete cytogenetic response
Time to reach MMR after restarting imatinib | Through study completion (five years)
  Time measured from the date of the reestart of imatinib until the achievement of MMR, days
Overall survival after imatinib discontinuation | Through study completion (five years)
  Overall survival is calculated from the date of imatinib discontinuation until the date of death by any cause
Progression-free survival after imatinib discontinuation | Through study completion (five years)
  PFS is calculated from the date of imatinib discontinuatio until the date of progression of the disease
Event-free survival after imatinib discontinuation | Through study completion (five years)
  Event-free is calculated from the date of imatinib discontinuation until the date of loss of complete hematologic response, disease progression or death
Molecular relapse free survival | Through study completion (five years)
  Calculated from the date of imatinib discontinuation until de loss of major molecular response

CONTACTS AND LOCATIONS:
Overall Officials: Katia B Pagnano, MD, Principal Investigator — University of Campinas
Locations (1):
- Centro de Hematologia e Hemoterapia - Universidade Estadual de Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for other researchers upon reasonable request with the principal investigator (Katia Pagnano) (all collected IPD, all IPD that underlie results in a publication)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available when summary data are published or otherwise made available
Access Criteria: The requests will be reviewed by the principal investigator Katia Pagnano and contacts should be done by email (kborgia@unicamp.br)
URL: https://www.hemocentro.unicamp.br/

REFERENCES:
- [Background] Gambacorti-Passerini C, Antolini L, Mahon FX, Guilhot F, Deininger M, Fava C, Nagler A, Della Casa CM, Morra E, Abruzzese E, D'Emilio A, Stagno F, le Coutre P, Hurtado-Monroy R, Santini V, Martino B, Pane F, Piccin A, Giraldo P, Assouline S, Durosinmi MA, Leeksma O, Pogliani EM, Puttini M, Jang E, Reiffers J, Piazza R, Valsecchi MG, Kim DW. Multicenter independent assessment of outcomes in chronic myeloid leukemia patients treated with imatinib. J Natl Cancer Inst. 2011 Apr 6;103(7):553-61. doi: 10.1093/jnci/djr060. Epub 2011 Mar 21. PMID 21422402
- [Background] Experts in Chronic Myeloid Leukemia. The price of drugs for chronic myeloid leukemia (CML) is a reflection of the unsustainable prices of cancer drugs: from the perspective of a large group of CML experts. Blood. 2013 May 30;121(22):4439-42. doi: 10.1182/blood-2013-03-490003. Epub 2013 Apr 25. PMID 23620577
- [Background] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Background] Rousselot P, Huguet F, Rea D, Legros L, Cayuela JM, Maarek O, Blanchet O, Marit G, Gluckman E, Reiffers J, Gardembas M, Mahon FX. Imatinib mesylate discontinuation in patients with chronic myelogenous leukemia in complete molecular remission for more than 2 years. Blood. 2007 Jan 1;109(1):58-60. doi: 10.1182/blood-2006-03-011239. Epub 2006 Sep 14. PMID 16973963
- [Background] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Bartley PA, Slader C, Field C, Dang P, Filshie RJ, Mills AK, Grigg AP, Melo JV, Hughes TP. Patients with chronic myeloid leukemia who maintain a complete molecular response after stopping imatinib treatment have evidence of persistent leukemia by DNA PCR. Leukemia. 2010 Oct;24(10):1719-24. doi: 10.1038/leu.2010.185. Epub 2010 Sep 2. PMID 20811403
- [Background] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Yeung DT, Dang P, Goyne JM, Slader C, Filshie RJ, Mills AK, Melo JV, White DL, Grigg AP, Hughes TP. Safety and efficacy of imatinib cessation for CML patients with stable undetectable minimal residual disease: results from the TWISTER study. Blood. 2013 Jul 25;122(4):515-22. doi: 10.1182/blood-2013-02-483750. Epub 2013 May 23. PMID 23704092
- [Background] Takahashi N, Kyo T, Maeda Y, Sugihara T, Usuki K, Kawaguchi T, Usui N, Okamoto S, Ohe Y, Ohtake S, Kitamura K, Yamamoto M, Teshima H, Motoji T, Tamaki T, Sawada K, Ohyashiki K. Discontinuation of imatinib in Japanese patients with chronic myeloid leukemia. Haematologica. 2012 Jun;97(6):903-6. doi: 10.3324/haematol.2011.056853. Epub 2011 Dec 16. PMID 22180435
- [Background] Cross NC, White HE, Muller MC, Saglio G, Hochhaus A. Standardized definitions of molecular response in chronic myeloid leukemia. Leukemia. 2012 Oct;26(10):2172-5. doi: 10.1038/leu.2012.104. Epub 2012 Apr 16. PMID 22504141
- [Background] Rousselot P, Charbonnier A, Cony-Makhoul P, Agape P, Nicolini FE, Varet B, Gardembas M, Etienne G, Rea D, Roy L, Escoffre-Barbe M, Guerci-Bresler A, Tulliez M, Prost S, Spentchian M, Cayuela JM, Reiffers J, Chomel JC, Turhan A, Guilhot J, Guilhot F, Mahon FX. Loss of major molecular response as a trigger for restarting tyrosine kinase inhibitor therapy in patients with chronic-phase chronic myelogenous leukemia who have stopped imatinib after durable undetectable disease. J Clin Oncol. 2014 Feb 10;32(5):424-30. doi: 10.1200/JCO.2012.48.5797. Epub 2013 Dec 9. PMID 24323036
- [Background] Yhim HY, Lee NR, Song EK, Yim CY, Jeon SY, Shin S, Kim JA, Kim HS, Cho EH, Kwak JY. Imatinib mesylate discontinuation in patients with chronic myeloid leukemia who have received front-line imatinib mesylate therapy and achieved complete molecular response. Leuk Res. 2012 Jun;36(6):689-93. doi: 10.1016/j.leukres.2012.02.011. Epub 2012 Mar 5. PMID 22398220
- [Background] Branford S, Yeung DT, Ross DM, Prime JA, Field CR, Altamura HK, Yeoman AL, Georgievski J, Jamison BA, Phillis S, Sullivan B, Briggs NE, Hertzberg M, Seymour JF, Reynolds J, Hughes TP. Early molecular response and female sex strongly predict stable undetectable BCR-ABL1, the criteria for imatinib discontinuation in patients with CML. Blood. 2013 May 9;121(19):3818-24. doi: 10.1182/blood-2012-10-462291. Epub 2013 Mar 20. PMID 23515925
- [Background] Falchi L, Kantarjian HM, Wang X, Verma D, Quintas-Cardama A, O'Brien S, Jabbour EJ, Ravandi-Kashani F, Borthakur G, Garcia-Manero G, Verstovsek S, Burger JA, Luthra R, Cortes JE. Significance of deeper molecular responses in patients with chronic myeloid leukemia in early chronic phase treated with tyrosine kinase inhibitors. Am J Hematol. 2013 Dec;88(12):1024-9. doi: 10.1002/ajh.23560. Epub 2013 Sep 12. PMID 23913852
- [Background] Rea D, Rousselot P, Guilhot J, Guilhot F, Mahon FX. Curing chronic myeloid leukemia. Curr Hematol Malig Rep. 2012 Jun;7(2):103-8. doi: 10.1007/s11899-012-0117-2. PMID 22410764
- [Background] Prost S, Relouzat F, Spentchian M, Ouzegdouh Y, Saliba J, Massonnet G, Beressi JP, Verhoeyen E, Raggueneau V, Maneglier B, Castaigne S, Chomienne C, Chretien S, Rousselot P, Leboulch P. Erosion of the chronic myeloid leukaemia stem cell pool by PPARgamma agonists. Nature. 2015 Sep 17;525(7569):380-3. doi: 10.1038/nature15248. Epub 2015 Sep 2. PMID 26331539
- [Background] Wang T, Xu J, Yu X, Yang R, Han ZC. Peroxisome proliferator-activated receptor gamma in malignant diseases. Crit Rev Oncol Hematol. 2006 Apr;58(1):1-14. doi: 10.1016/j.critrevonc.2005.08.011. Epub 2006 Jan 18. PMID 16388966